CLINICAL TRIAL: NCT03753776
Title: Phase III Trial Evaluating Radium Bromatum Homeopathic Treatment Efficacy on Radiodermatitis Prevention and Treatment for Breast Cancer Women
Acronym: HOMEORAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0601; 2018-002406-32 (EudraCT Number)
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Homeopathy; Radium bromatum; Apis mellifica; Belladonna; Radiodermatitis; Radiotherapy; Prevention; Treatment; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: A first randomization will establish two groups : placebo versus homeopathy (Radium bromatum), and if patients develop a radiodermatitis of grade 2 or higher, a second randomization will take place, with two groups : placebo versus homeopathy (Radium bromatum, Apis mellifica, and Belladonna)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither patients receiving pills nor doctors evaluating radiodermatitis know the nature of treatment (placebo or homeopathy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Radium bromatum placebo group (Placebo Comparator): Placebo group will receive placebo pills of Radium bromatum during radiotherapy
  Interventions: Drug: Placebo pills of Radium bromatum
- Radium bromatum group (Experimental): Radium bromatum group will receive homeopathic Radium bromatum pills during radiotherapy
  Interventions: Drug: Radium bromatum pills
- Radium bromatum/Apis mellifica/Belladonna placebo group (Placebo Comparator): Placebo group will receive Radium bromatum/Apis mellifica/Belladonna placebo pills to treat grade 2 or higher radiodermatitis
  Interventions: Drug: Radium bromatum/Apis mellifica/Belladonna placebo pills
- Radium bromatum/Apis mellifica/Belladonna group (Experimental): Radium bromatum/Apis mellifica/Belladonna group will receive homeopathic Radium bromatum/Apis mellifica/Belladonna pills to treat grade 2 or higher radiodermatitis
  Interventions: Drug: Radium bromatum/Apis mellifica/Belladonna pills

INTERVENTIONS:
Drug: Placebo pills of Radium bromatum — Placebo pills of Radium bromatum will be taken since 48h before radiotherapy and until 15 days after the end of radiation, or until grade 2 or higher radiodermatitis apparition
  Other Names: Radium bromatum placebo
  Arms: Radium bromatum placebo group
Drug: Radium bromatum pills — Homeopathic Radium bromatum pills will be taken since 48h before radiotherapy and until 15 days after the end of radiation, or until grade 2 or higher radiodermatitis apparition
  Other Names: Radium bromatum
  Arms: Radium bromatum group
Drug: Radium bromatum/Apis mellifica/Belladonna placebo pills — Placebo pills of Radium bromatum, Apis mellifica and Belladonna will be taken since grade 2 or higher radiodermatitis and until 15 days after the end of radiation
  Other Names: Radium bromatum/Apis mellifica/Belladonna placebo
  Arms: Radium bromatum/Apis mellifica/Belladonna placebo group
Drug: Radium bromatum/Apis mellifica/Belladonna pills — Pills of Radium bromatum, Apis mellifica and Belladonna will be taken since grade 2 or higher radiodermatitis and until 15 days after the end of radiation
  Other Names: Radium bromatum/Apis mellifica/Belladonna
  Arms: Radium bromatum/Apis mellifica/Belladonna group

SUMMARY:
Breast cancer is the second most frequent cancer worldwide. Principal therapy consists in radiotherapy, but this technic has sides effects as radiodermatitis, concerning about 90 percent of women treated.

Risk of flushing could be reduced by hygienic rules, but no treatment proved its efficacy to prevent radiodermatitis.

Homeopathy is popular but also contested. No clinical trial proved its efficacy for this indication. The present study aims at evaluating Radium bromatum efficacy (homeopathy), compared to placebo, to prevent radiodermatitis apparition for women treated for breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the second most frequent cancer worldwide, and the most frequent in France. Principal therapy consists in radiotherapy, that is locoregional, using radiations to kill cancerous cells.

Radiotherapy has sides effects as radiodermatitis, concerning about 90 percent of women treated. Radiodermatitis could be described with three factors : redness, heat, and edema.

Risk of flushing could be reduced by hygienic rules concerning hydratation, clothes, and toilet.

Nowadays, no treatment proved homeopathic efficacy to prevent radiodermatitis. This treatment is popular but also contested. No clinical trial proved its efficacy for this indication. The present study aims at evaluating Radium bromatum efficacy (homeopathy), compared to placebo, to prevent radiodermatitis apparition for women treated for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Major patient;
* Indication of curative intent radiotherapy for breast cancer treated with conservative treatment. Accepted radiotherapy scheme: 50 Gy (main) + 16 Gy on the tumor bed (additional dose);
* Patient affiliated or entitled to a social security scheme;
* Patient who signed an informed consent form.

Exclusion Criteria:

* Pregnant or lactating woman;
* Legal incapacity or limited legal capacity. Medical or psychological conditions that do not allow the subject to understand the study and sign the consent
* Patient followed by a liberal homeopath;
* Patient with bilateral breast cancer;
* Patient with in situ breast cancer;
* Patient with known cognitive impairment;
* Patient with known allergy and / or intolerance and / or malabsorption to fructose, glucose, galactose;
* Patient with a known deficiency in sucrase / isomaltase / lactase.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Percentage diminution of grade 2 or higher radiodermatitis in Radium bromatum group | Week 6
  Percentage diminution of grade 2 or higher radiodermatitis in Radium bromatum group will be measure with the RTOG (Radiation Therapy Oncology Group) scale. A diminution of 10% between Radium bromatum group and placebo group will be considered as significant

SECONDARY OUTCOMES:
Radiodermatitis frequency | Week 6
  Number of Radiodermatitis according to the RTOG (Radiation Therapy Oncology Group) scale will be reported.
Radiodermatitis duration | Week 6
  Radiodermatitis duration will be reported in days.
Radiodermatitis delays | Week 6
  Radiodermatitis delays will be reported in days.
Number of concomitant treatments | Week 6
  Number of concomitant treatments will be reported.
Pain measure | Week 6
  Measure of pain will be reported, calculated with a oral scale between 0 and 10.
Level of Quality of life | Week 6
  Level of Quality of life will be measured between 0 to 100 with the EQ-5D questionnaire (european quality of life number 5)
Satisfaction measure | Week 6
  Satisfaction will be measured with a oral scale between 0 (no satisfaction) and 3 (full satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Beneton, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No